CLINICAL TRIAL: NCT02836886
Title: Searching for Oncogenic Viruses in Sézary Cells Using a Novel Viral Discovery Technique, VirCapSeq-VERT
Brief Title: VircapSeq Virus Detection in Sézary Syndrome
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAQ9017
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Sézary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Sezary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample: two tubes collected by standard blood draw (venipuncture) procedure. The total amount of blood drawn will be about two teaspoons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sézary syndrome: Patients diagnosed with Sézary syndrome diagnosed according to the WHO-EORTC criteria.

SUMMARY:
This study will be using this technique, called "VirCapSeq-VERT" to analyze the white blood cells of patients with Sézary syndrome. This could provide the foundation for future studies looking to understand the role that viruses play in the origin of Sézary syndrome. This could have important implications for the future development of new and effective therapies for the disease.

DETAILED DESCRIPTION:
Cutaneous T-cell lymphoma (CTCL) is a rare lymphoproliferative disorder characterized by malignant CD4+ T-cells that infiltrate the skin. While most cases are confined to skin, CTCL is also capable of affecting the blood, lymph nodes, and visceral organs. Sézary Syndrome (SS) is a leukemic variant of the disease with a poor prognosis and can arise with or without cutaneous involvement. The pathogenesis of CTCL is poorly understood, but chronic antigen stimulation possibly due to a bacterial or viral infection or colonization of the skin may lead to malignant transformation of the skin resident T cells. Colonization of the skin of CTCL patients with Staphylococcus aureus is common and can lead to the clonal expansion of malignant T cells in the skin. However, its role as an etiological agent is unlikely, considering commonality of S.aureus and rarity of the skin T-cell lymphomas. Mounting evidence suggests that oncogenic viral pathogen may play a role, but all efforts to implicate certain viruses, such as retroviruses or herpesviruses have yielded inconsistent results. This study will use the most sensitive method to date, a novel viral detection technique capable of detecting every known vertebrate virus in tissue samples, called "Virome Capture Sequencing Platform for Vertebrate Viruses (VirCapSeq-VERT)." This allows it to detect previously undiscovered viruses that diverge from known sequences by as much as 40%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Sézary syndrome diagnosed according to the WHO-EORTC classification.

Exclusion Criteria:

* Pregnant patients.
* Patients with known anemia with documented <7.5 mg/dL.
* Patients who are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Sézary syndrome diagnosed according to the WHO-EORTC criteria.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larisa G Geskin, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willemze R, Jaffe ES, Burg G, Cerroni L, Berti E, Swerdlow SH, Ralfkiaer E, Chimenti S, Diaz-Perez JL, Duncan LM, Grange F, Harris NL, Kempf W, Kerl H, Kurrer M, Knobler R, Pimpinelli N, Sander C, Santucci M, Sterry W, Vermeer MH, Wechsler J, Whittaker S, Meijer CJ. WHO-EORTC classification for cutaneous lymphomas. Blood. 2005 May 15;105(10):3768-85. doi: 10.1182/blood-2004-09-3502. Epub 2005 Feb 3. PMID 15692063
- [Background] Siegel RS, Pandolfino T, Guitart J, Rosen S, Kuzel TM. Primary cutaneous T-cell lymphoma: review and current concepts. J Clin Oncol. 2000 Aug;18(15):2908-25. doi: 10.1200/JCO.2000.18.15.2908. PMID 10920140
- [Background] Henn A, Michel L, Fite C, Deschamps L, Ortonne N, Ingen-Housz-Oro S, Marinho E, Beylot-Barry M, Bagot M, Laroche L, Crickx B, Maubec E. Sezary syndrome without erythroderma. J Am Acad Dermatol. 2015 Jun;72(6):1003-9.e1. doi: 10.1016/j.jaad.2014.11.015. PMID 25981000
- [Background] Lessin SR, Vowels BR, Rook AH. Retroviruses and cutaneous T-cell lymphoma. Dermatol Clin. 1994 Apr;12(2):243-53. PMID 8045036
- [Background] Willerslev-Olsen A, Krejsgaard T, Lindahl LM, Bonefeld CM, Wasik MA, Koralov SB, Geisler C, Kilian M, Iversen L, Woetmann A, Odum N. Bacterial toxins fuel disease progression in cutaneous T-cell lymphoma. Toxins (Basel). 2013 Aug 14;5(8):1402-21. doi: 10.3390/toxins5081402. PMID 23949004
- [Background] Mirvish JJ, Pomerantz RG, Falo LD Jr, Geskin LJ. Role of infectious agents in cutaneous T-cell lymphoma: facts and controversies. Clin Dermatol. 2013 Jul-Aug;31(4):423-431. doi: 10.1016/j.clindermatol.2013.01.009. PMID 23806159
- [Background] Briese T, Kapoor A, Mishra N, Jain K, Kumar A, Jabado OJ, Lipkin WI. Virome Capture Sequencing Enables Sensitive Viral Diagnosis and Comprehensive Virome Analysis. mBio. 2015 Sep 22;6(5):e01491-15. doi: 10.1128/mBio.01491-15. PMID 26396248
- [Background] Anderson ME, Nagy-Szakal D, Jain K, Patrone CC, Frattini MG, Lipkin WI, Geskin LJ. Highly Sensitive Virome Capture Sequencing Technique VirCapSeq-VERT Identifies Partial Noncoding Sequences but no Active Viral Infection in Cutaneous T-Cell Lymphoma. J Invest Dermatol. 2018 Jul;138(7):1671-1673. doi: 10.1016/j.jid.2018.01.024. Epub 2018 Feb 7. No abstract available. PMID 29427587

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sézary Syndrome
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sézary Syndrome
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 65 [58 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Viral Sequences Present in Malignant T Cells of Patients With Sézary Syndrome
Time Frame: Through study completion, an average of 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sézary Syndrome
Number analyzed (Participants) | 6
Participants | 6

2. Other Pre Specified Outcome: Number of Coding Sequences for Viral Pathogens Extracted From T Cells of Patients With Sézary Syndrome
Time Frame: Through study completion, an average of 4 months
Measure: Number; unit: coding sequences for viral pathogens
Arm/Group | Sézary Syndrome
Number analyzed (Participants) | 6
coding sequences for viral pathogens | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 months
Arm/Group | Sézary Syndrome
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No